CLINICAL TRIAL: NCT07150962
Title: A Phase I Clinical Study Comparing the Relative Bioavailability, Safety and Tolerability of the First-generation and Second-generation Formulations of HRS9531 Tablets and Exploring the Safety, Tolerability and Pharmacokinetic Characteristics of Single-dose Escalation of the Second-generation Formulation
Brief Title: Relative Bioavailability of First vs Second-Generation Formulations of HRS9531 Tablets in Obese or Overweight Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Fujian Shengdi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRS9531-T-103
Record Dates: First submitted 2025-08-27; First posted 2025-09-02 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: Overweight or Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multiple ascending dose group (Experimental)
  Interventions: Drug: HRS-9531 Tablet
- Single ascending dose group (Experimental)
  Interventions: Drug: HRS-9531 Tablet

INTERVENTIONS:
Drug: HRS-9531 Tablet — HRS-9531 tablet.

SUMMARY:
This study aims to compare the relative bioavailability, safety and tolerability of the first-generation and second-generation formulations of HRS9531 tablets, as well as to explore the safety, tolerability and pharmacokinetic characteristics of the second-generation formulation in terms of single-dose escalation.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand the trial procedures and possible adverse events, be able and willing to provide a written informed consent;
2. Male subjects aged 18-55 years on the date of signing informed consent (inclusive);
3. Body weight ≥65 kg, body mass index (BMI) within the range of 24.0-35.0 kg/m2 (inclusive);
4. The weight change within the previous 3 months should not exceed 5 kilograms.
5. Based on the patient's past medical history, physical examination, vital signs, laboratory tests and electrocardiogram (ECG) examinations, the researchers determined that the overall overweight and obese subjects were included.

Exclusion Criteria:

1. Those who are known or suspected to be allergic to any component of the investigational drug or related products; or those who have a history of multiple or severe allergies to drugs or foods, or a history of severe immediate allergic reactions;
2. Chronic or severe medical history of the respiratory system, circulatory system, digestive system, urinary system, blood system, endocrine system, immune system, nervous system, mental system, etc., or those with existing systemic diseases mentioned above, and judged by the investigator to be unsuitable to participate in this study;
3. Having a history of hypertension or when the researchers determine during the screening that the blood pressure is abnormal and has clinical significance;
4. Those with a history of obvious gastrointestinal diseases or related symptoms (such as nausea, vomiting, heartburn sensation or diarrhea), conditions that affect gastric emptying (such as pyloric stenosis), or who have undergone any gastrointestinal surgery (such as weight loss surgery; except for intestinal polyp resection and appendectomy), or who had acute diarrhea within the previous 7 days; diarrhea is defined as watery stools and/or more than 3 bowel movements per day;
5. Participation in clinical trials of any drug or medical device in the 3 months or 5 half-lives, whichever longer, prior to dosing;
6. Blood donation history or blood loss ≥400 mL within 3 months or ≥200 mL within 1 month before dosing, or received blood transfusion within 3 months before dosing;
7. Hepatitis B surface antigen (HBsAg), HIV antibody, hepatitis C virus antibody (HCVAb), treponema pallidum specific antibody detection, positive;
8. Those who have a history of drug abuse or drug use, or who have a positive result in the urine drug screening test during the screening period;
9. Heavy drinkers (average weekly alcohol consumption of ≥ 14 units in the six months prior to screening: 1 unit of beer = 285 mL, or spirits = 25 mL, or wine = 100 mL; average daily smoking ≥ 5 cigarettes); those unable to quit smoking and drinking during the trial; those with positive alcohol blood tests.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 168 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Area under the curve from Time Zero to Time of last quantifiable concentration (AUCtau) | From Day 14 to Day 15.
Adverse event (AE) | Screening period up to Day 35.
Serious adverse event (SAE) | Screening period up to Day 35.

SECONDARY OUTCOMES:
The maximum plasma concentration (Cmax) | On the 35th day after continuous administration.
Time to maximum plasma concentration (Tmax) | On the 35th day after continuous administration.
Area under the concentration-time curve (AUC) | On the 35th day after continuous administration.
Time to maximum plasma concentration (Tmax) | Post-dose from Day 1 to Day 183.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Undecided